CLINICAL TRIAL: NCT02590042
Title: A Phase I Open-labeled, Single-arm, Single-centred Study to Test the Safety of ADSC-SVF-002 in Subjects With Soft Tissue Defects or Abnormal Wound Healing
Brief Title: Safety of Adipose-Derived Stem Cell Stromal Vascular Fraction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AdiSave Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJS-CT-001
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Abnormally Healing Wounds; Scars; Soft Tissue Defects
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADSC-SVF-002 (Experimental): Cells will be administered at 1x10^6 cells/mL of defect. If administered with fat, the cells will be administered at 1.2x10^6 cells/mL of defect.
  Interventions: Biological: ADSC-SVF-002

INTERVENTIONS:
Biological: ADSC-SVF-002 — ADSC-SVF with the following identity:
  Less than or equal to 10% each CD34 and CD45 positive cells At least 70% each CD90, CD73 and CD105 positive cells Viability of at least 85% Mean Florescence Intensity of less than or equal to 100 C12FDG 0-5-2.5x10^6 cells/g of liposuctioned (hydrated fat)
  Other Names: ADSC-SVF manufactured by AdiSave

SUMMARY:
A single-arm, open-labeled, single-center, descriptive and exploratory safety trial using ADSC-SVF-002. ADSC-SVF-002 is an autologous adipose derived stem cell (ADSC)-containing stromal vascular fraction (SVF) obtained from subcutaneous fat harvested by liposuction from a patient. As a cellular therapy product, ADSC-SVF-002 (fresh or cryopreserved) will be administered subcutaneously via injection, with or without unprocessed autologous fat (fresh or cryopreserved), into soft tissue defects and abnormally healing wounds. The primary objective of the trial is to demonstrate the safety of ADSC-SVF-002 in a population of subjects with soft tissue defects or abnormal wound healing who are still symptomatic despite being managed by conventional therapies.

DETAILED DESCRIPTION:
Protocol Number: SJS-CT-001 Phase: Pilot study Methodology: Open label, single-arm Study Duration: Six months after accrual and treatment of the last patient Study Center(s): Single-center Objectives: To demonstrate the safety of subcutaneous administration of autologous ADSC-SVF-002 in a population of subjects with soft tissue defects or abnormal wound healing who are still symptomatic despite being managed by conventional therapies.

Number of Subjects: 10 Diagnosis and Main Inclusion Criteria: Subject has soft tissue deficiencies, soft tissue post traumatic malformations, scars, and/or abnormal wound healing.

Study Product, Dose, Route, Regimen: ADSC-SVF-002. 1.0x106 cells/mL defect (when administered without fat) to 1.2x106 cells/mL defect (when administered with fat). Subcutaneous injection.

Duration of administration: Administration of the product takes approximately 30 minutes. Administered once.

Reference therapy: N/A

Statistical Methodology: Safety outcomes will be reported with descriptive statistics. Secondary (efficacy) outcomes will be assessed relative to baseline (screening) as follows:

* For outcomes assessed at multiple follow-up visits, one-way ANOVAs followed by the Tukey's test will be conducted
* For outcomes assessed at one follow-up visit, a Student's t-test will be conducted.

Data will be reported as mean ± SD and p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has soft tissue deficiencies, soft tissue post traumatic malformations, scars, and/or abnormal wound healing.
2. Subject is an adult male or non-pregnant female between the ages of 18 to 80 years.
3. Subject is able to undergo a liposuction procedure in the opinion of the investigator or per facility guidelines.
4. Subject is able to read, understand and sign a written Informed Consent to participate in the study.
5. Subject is willing and able to comply with the study protocol, including requirements for taking and abstaining from medications.

Exclusion Criteria:

1. The subject is a woman of child-bearing potential (not surgically sterile or post-menopausal for at least 1 year as documented in medical history), but is not using a highly effective method of contraception [oral, injected or implanted hormonal methods of contraception; intrauterine device (IUD) or intrauterine system (IUS); condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; or male sterilization (vasectomy)].
2. Subject has a history of cancer and/or any known conditions/diseases prone to malignancy.
3. Subject has significant cardiac, renal, or hepatic failure or any other disease that may interfere with the ability to interpret the results of the study.
4. Subject has an infection, cellulitis, or osteomyelitis diagnosed by MRI and microbiologic culture results.
5. Subject has an autoimmune disorder.
6. Subject has a connective, metabolic or atrophic skin disease.
7. Subject is under chronic anticoagulant therapy.
8. Subject has a Body Mass Index (BMI) >30.
9. Subject is positive for HBs antigen, HCV antibody, or HIV antibody.
10. Subject has received other investigational drug/drugs or unapproved medication within 3 months before registration in this study.
11. Subject has a history of hematopoietic stem cell transplantation or radio immunotherapy.
12. Subject has a recent and significant weight loss, the cause of which has not been determined.
13. Subject has a history of hereditary linked malignancy in a first-degree relative (parent, child, sibling).
14. Subject is participating in another clinical trial within 6 weeks prior to registration in this study.
15. Subject has a psychiatric disorder that in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Continuous monitoring of safety via laboratory tests and physical examinations | Screening, 48 hours after procedure, and at post-treatment months 1, 2 and 6
  Continuous monitoring of safety as requested by Health Canada

SECONDARY OUTCOMES:
Physician satisfaction with wound cosmesis, assessed using the Hollander Wound Evaluation Scale | Screening, 48 hours after procedure, and at post-treatment day 10 and months 1-6
Patient satisfaction with wound cosmesis, assessed using the 100 mm vertical line visual analogue scale | Screening, 48 hours after procedure, and at post-treatment day 10 and months 1-6

CONTACTS AND LOCATIONS:
Overall Officials: Sarah HM Wong, MD, Principal Investigator — Forest Hill Institute of Aesthetic Plastic Surgery
Locations (1):
- Forest Hill Institute of Aesthetic Plastic Surgery, Toronto, Ontario, Canada